CLINICAL TRIAL: NCT01898429
Title: Deep Brain Stimulation for Treatment-Resistant Depression
Brief Title: Deep Brain Stimulation (DBS) for Treatment-Resistant Depression (TRD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Holtzheimer (Other)
Responsible Party: Sponsor-Investigator, Paul Holtzheimer, Deputy Director for Research at the National Center for PTSD, Associate Professor for Dartmouth/Dartmouth Hitchcock., Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D12051; 23293 (Other: Dartmouth Committee for the Protection of Human Subjects)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Treatment Resistant Depression; Depressive Disorder, Treatment-Resistant; Depression, Bipolar
Keywords: Treatment Resistant Depression; Treatment Refractory Depression; Treatment Resistant Bipolar Disorder; Treatment Refractory Bipolar Disorder; Deep brain stimulation; DBS
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Bipolar Disorder | interventions — Deep Brain Stimulation; Drug Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left-sided SCC DBS (Active Comparator): Active Stimulation of the left-sided electrode
  Interventions: Device: SCC DBS
- Right-sided SCC DBS (Active Comparator): Active stimulation of the right-sided electrode
  Interventions: Device: SCC DBS

INTERVENTIONS:
Device: SCC DBS — Deep Brain Stimulator
  Other Names: Libra(TM) Implantable Deep Brain Stimulation (DBS) System

SUMMARY:
In this pilot study, we propose to test whether high frequency stimulation of the subcallosal cingulate (SCC) is a safe and efficacious antidepressant treatment in five TRD patients, to compare the effects of left-sided vs. right-sided stimulation, and to investigate potential mechanisms of action of this intervention. Importantly, this study will be used to assess the need for and assist in planning a larger, more definitive trial of SCC DBS for TRD.

DETAILED DESCRIPTION:
The U.S. lifetime prevalence of major depressive disorder (MDD) is 17%. A number of treatments are available for depression including medications, psychotherapy and various somatic treatments. Unfortunately, up to two-thirds of patients remain symptomatic following first-line treatment and a third fail to achieve remission (defined as full resolution of depressive symptoms) after four established treatments; approximately 10%-20% of depressed patients may show virtually no improvement despite multiple, often aggressive treatments. Thus, a conservative estimate places the U.S. prevalence of treatment-resistant depression (TRD) at 1%-3%. TRD has a high risk of suicide, is a major cause of disability and is responsible for doubling of overall health care costs.

For patients with TRD there are limited evidence-based treatment options. Transcranial magnetic stimulation (TMS) may have efficacy for patients that have failed no more than one antidepressant medication 10-12, but response and remission rates are relatively low (under 30% and 20% respectively). Vagus nerve stimulation (VNS) may have efficacy in patients that have failed 4-6 antidepressant treatments but long-term response and remission rates are again low (about 20% and 10% respectively). Electroconvulsive therapy(ECT) can be effective in TRD patients with remission rates of 50%-60%. However, more than 70% of TRD patients will relapse within 6 months following a successful acute treatment course. For patients that have failed ECT, there are no evidence-based treatment options. Therefore, there is great need for novel treatment approaches for TRD.

Prior clinical trials have shown that SCC DBS has the potential to be a valuable treatment option for patients with TRD. Further developing this treatment will involve confirming its effectiveness and identifying ways to optimize its use. In this study we intend to test the safety and efficacy of chronic SCC DBS as a treatment for TRD and compare the safety and efficacy of left-sided versus right-sided stimulation using a double-blind, randomized, cross-over design.

ELIGIBILITY:
A partial list of eligibility criteria includes:

* Age 18-70 years old
* Ability to provide written informed consent
* Current Major Depressive Episode (MDE), secondary to either Major Depressive Disorder or Bipolar Disorder (I, II or NOS)
* A current depressive episode of at least 12 months duration
* For patients with a bipolar disorder, the last hypomanic or manic episode must have been at least 2 years before study entry
* A maximum Global Assessment of Functioning of 50
* Able to tolerate general anesthesia, DBS surgery and MRI scans
* No significant cerebrovascular risk factors or a previous stroke, documented major head trauma or neurodegenerative disorder
* No currently active clinically significant Axis I psychiatric diagnosis or a personality disorder likely to interfere with the study
* No evidence of global cognitive impairment
* Lives locally or willing to relocate to the area for up to One Year

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Holtzheimer, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in Jan 2012. Participants were enrolled from July 2013 through January 2016. Patients were primarily recruited by clinicaltrials.gov and through information provided to providers.
Pre-assignment Details: All participants entered the left unilateral stimulation phase first; all then transitioned to the right side. This decision was made by the unblinded programmer. Patients and raters were still blinded to treatment allocation.
Groups:
- Bilateral SCC DBS: 12 weeks of bilateral SCC DBS
Period: Phase 1
Arm/Group | Left-sided SCC DBS | Right-sided SCC DBS | Bilateral SCC DBS
Started | 5 | 0 | 0
Completed | 5 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2
Arm/Group | Left-sided SCC DBS | Right-sided SCC DBS | Bilateral SCC DBS
Started | 0 | 5 | 0
Completed | 0 | 5 | 0
Not Completed | 0 | 0 | 0
Period: Phase 3
Arm/Group | Left-sided SCC DBS | Right-sided SCC DBS | Bilateral SCC DBS
Started | 0 | 0 | 5
Completed | 0 | 0 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients entered the left-sided phase first, then crossed over to the right-sided phase.
Groups:
- All Participants: Active Stimulation of the left-sided electrode in the first phase (followed by right-sided stimulation in the second phase)
  SCC DBS: Deep Brain Stimulator
Arm/Group | All Participants
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Hamilton Depression Rating Scale (17 items) [Mean (Standard Deviation); unit: units on a scale] — Standard rating scale for depression severity. Administered by a rater trained and tested for interrater reliability.
  units on a scale | 22.4 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of 12 Weeks of Left Unilateral DBS vs. 12 Weeks Right Unilateral DBS on Change in 17-item Hamilton Depression Rating Scale (HDRS-17)
Description: Baseline HDRS-17 is defined as the average of 4 weekly HDRS-17 in the 4 weeks leading up to surgery. Change in HDRS-17 after 12 weeks of left-sided stimulation (compared to baseline) will be compared to change in HDRS-17 after 12 weeks of right-sided stimulation (compared to baseline). The scale ranges from 0-48 with higher scored indicating more severe depression. A cutoff of 7 or below is considered remission from depression. A decrease of at least 50% from baseline is considered an antidepressant response.
Time Frame: baseline, 12 weeks of phase 1, 12 weeks of phase 2 and 12 weeks of phase 3 (bilateral stimulation)
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 5
units on a scale
  Baseline | 22.35 [20.25 to 25.50]
  12 weeks left-sided stimulation | 18.8 [16 to 20]
  12 weeks right-sided stimulation | 21.4 [18 to 25]
  12 weeks of bilateral stimulation | 17.4 [6 to 22]

ADVERSE EVENTS:
Time Frame: 40 weeks following surgery to implant the DBS device
Description: adverse events data were collected using the SAFTEE developed by the NIH
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=5)
altered mental status (Nervous system disorders) | 1 (1) — confusion related to oxycodone use post-surgery leading to emergency room visit (no hospitalization required)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=5)
multiple (General disorders) | 5 (38) — Multiple mild adverse events were identified using the SAFTEE. Only 1 of 38 (pain at the IPG implantation site) was deemed to be related to the surgery or study device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes